CLINICAL TRIAL: NCT06721052
Title: Retrospective Evaluation of Ultrasound-guided Deep Iliacus Plane Block / Meta-PENG: Another Novel Fascial Plane Block
Brief Title: Retrospective Evaluation of Efficacy of Meta-PENG Block
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Other Study IDs: Medipol Hospital 39
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hip Fractures; Hip Injuries
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group meta-PENG block: We performed meta-PENG block in patients who underwent hip surgery under spinal or general anesthesia
  Interventions: Drug: meta-Peng block; Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: meta-Peng block — The convex transducer was positioned obliquely in a superolateral to inferomedial direction just above the femoral crest. Anatomical structures including AIIS, iliopubic eminence, sartorius muscle, iliopsoas muscle, psoas tendon, artery, vein, and iliac fascia were identified sono-anatomically. The AIIS was centered in the transducer image. To determine the insertion point of the rectus femoris tendon (RFT) on the AIIS, the transducer was rotated sagittally, and the level where the RFT ends cephalically was identified. After identifying the target, the transducer was obliquated again to visualize the IPE. The 22G x 100 mm block needle was advanced in-plane from lateral to inferomedial towards the potential space between the IPM and AIIS. After confirming the target plane with a few mL of saline, 30-40 mL of 0.25% bupivacain was applied to the area. The spread of injectate was observed beneath the IPM, below the psoas tendon, and around the iliacus muscle within the iliac fascia.
Drug: Postoperative analgesia management — We ordered 400 mg intravenous ibuprofen for the patients every 8 hours during the postoperative period. We planned to perform 100 mg tramadol as a rescue analgesic if the patient's NRS score was above 4. We observed the patients for 24 hours in the postoperative period.

SUMMARY:
The components of the lumbar plexus and capture the articular branches of hip capsule may be effectively blocked by administering a relatively high volume of local anesthetic deep to the iliacus muscle at the level of the anterior inferior iliac spine. We can provide both the blockade of the pericapsular nerve group supplying the hip capsule and the cutaneous blockade. Here, we aimed to present our novel technique we named 'deep iliacus plane block (DIPB)'.

DETAILED DESCRIPTION:
Many regional anesthesia techniques are used in hip surgeries for various goals, such as optimizing neuraxial positioning and relieving pain in the perioperative period, and have been the subject of clinical researches in the last few decades.

The lumbar plexus is important in administering anesthesia and analgesia during hip and knee surgeries. Comprising the femoral nerve (FN), lateral femoral cutaneous nerve (LFCN), and obturator nerve, it collaborates with the sacral plexus to ensure comprehensive innervation of the lower limb.

We hypothesized that by administering a relatively high volume of local anesthetic deep to the iliacus muscle at the level of the anterior inferior iliac spine (AIIS), we could effectively block the lumbar plexus components and capture the hip capsule's articular branches. We can ensure both the blockade of the pericapsular nerve group supplying the hip capsule and the cutaneous blockade. Here, we aimed to present our cadaveric evaluation and retrospective evaluation of patients underwent meta-PENG block, which we consider the proof-of-concept for our hypothesis of the technique we named 'deep iliacus plane block (DIPB)'.

ELIGIBILITY:
Inclusion Criteria:

* ASA-1, ASA-2 and ASA-3 patients who underwent hip surgery under spinal or general anesthesia

Exclusion Criteria:

Anticoagulant drug use Known allergy to the medications to be used Infection in the area where the needle will be inserted Missing data

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent hip fracture surgery due to fracture or another reason
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Pain scores (Numerical rating scale-NRS) | Before block, 30 min after block
  Comparison of NRS before block, after block, and during position for surgery
Pain scores (Numerical rating scale-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, and 24 hours
  The primary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded

SECONDARY OUTCOMES:
Need for rescue analgesia (tramadol) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Pun M, Ng T, Vermeylen K, Tran J. Innervation of the hip joint: implications for regional anaesthesia and image-guided interventional pain procedures. BJA Educ. 2024 Jun;24(6):191-202. doi: 10.1016/j.bjae.2024.02.005. Epub 2024 Apr 8. No abstract available. PMID 38764441
- [Background] Vermeylen K, Soetens F, Leunen I, Hadzic A, Van Boxtael S, Pomes J, Prats-Galino A, Van de Velde M, Neyrinck A, Sala-Blanch X. The effect of the volume of supra-inguinal injected solution on the spread of the injectate under the fascia iliaca: a preliminary study. J Anesth. 2018 Dec;32(6):908-913. doi: 10.1007/s00540-018-2558-9. Epub 2018 Sep 24. PMID 30250982
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Nielsen ND, Madsen MN, Ostergaard HK, Bjorn S, Pedersen EM, Nielsen TD, Soballe K, Borglum J, Bendtsen TF. An iliopsoas plane block does not cause motor blockade-A blinded randomized volunteer trial. Acta Anaesthesiol Scand. 2020 Mar;64(3):368-377. doi: 10.1111/aas.13498. Epub 2019 Nov 13. PMID 31650529